CLINICAL TRIAL: NCT01356836
Title: The Association Between Different Monocyte Subsets and Coronary Collateral Development
Status: Completed | Type: Observational
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Türkiye Yüksek İhtisas Education and Research Hospital, Specialist of Cardiology
Other Study IDs: Monocyte subsets
Record Dates: First submitted 2011-05-17; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Artery Disease; Coronary Ischemia
Keywords: Coronary collateral development; monocyte subsets; collateralization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Good-poor collateral: Patients who had good and poor collaterals formed 2 groups
- Good collateral, Poor collateral

SUMMARY:
Collateral growth and coronary angiogenesis are chronic adaptations to myocardial ischemia. Collateralization helps to restore blood flow and as a result salvages myocardium in severely ischemic myocardial regions. Thus, good collateral development in patients with severe coronary artery disease (CAD) improves ventricular function and prognosis (1-3).

However, coronary collateral development is different among patients even with similar degrees of coronary artery stenosis. Several factors, such as diabetes mellitus (4) and duration of myocardial ischemic symptoms (5) have been reported to effect coronary collateral development. At the cellular level, inflammatory cells, especially monocytes have an important role in collateralization. In a series of experimental studies with animals, it has been shown that monocytes are important elements for development of collateral vessels (6-7). In a recent study, it has been demonstrated that increased circulating monocyte count is related to good collateral development in patients with stable coronary artery disease (8).

Monocytes in human blood are heterogeneous and can be classified into two subsets according to the presence or absence of the FcγRIII receptor CD16 (9): CD14++CD16- monocytes characterized by high level expression of the CD14 cell surface receptor but no expression of CD16 receptor, and CD14+CD16+ monocytes characterized by the co-expression of CD16 receptor with either high or low level expression of the CD14 receptor. These subsets differ in function and response to several cytokines.

Our aim in this study was to find out any possible relationship between the levels of circulating monocyte subsets and coronary collateral development.

ELIGIBILITY:
Inclusion Criteria:

* > 95% stenosis of at least one major coronary artery in their first coronary angiogram

Exclusion Criteria:

* previous percutaneous or surgical revascularization history
* evidence of ongoing infection and inflammation
* known malignancy and chronic kidney disease (serum creatinine > 1.5 mg/dl
* diabetic patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who were found to have >95% stenosis of at least one major coronary artery in their first coronary angiogram were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 1Türkiye Yüksek İhtisas Education and Research Hospital, Department of Cardiology, Ankara, Turkey (Türkiye)